CLINICAL TRIAL: NCT04297423
Title: Eficacia y Tolerabilidad de Dos Productos de Volumen Reducido Para la Colonoscopia de Cribado: Ensayo Comparativo Paralelo Aleatorizado
Brief Title: Two Low Volume Regimens for Colorectal Cancer Screening Colonoscopy
Acronym: LOWOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Casen Recordati S.L. (Industry); Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, María Pellisé, Principal Investigator. Attending physician Gastroenterology department., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2019/0872
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
Keywords: Bowel Preparation Solutions; Screening colonoscopy; Adenoma detection rate; Tolerability; 1L PEG plus ascorbate; Magnesium citrate plus picosulphate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: A comparative, parallel, randomized, non-inferiority, non-blinded, single-centre and low-intervention clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plenvu (Experimental): Plenvu split dose
  Interventions: Drug: Plenvu
- Citrafleet (Active Comparator): citrafleet in split dose
  Interventions: Drug: Plenvu

INTERVENTIONS:
Drug: Plenvu — randomization 1:1
  Other Names: citrafleet

SUMMARY:
Colorectal cancer is the first neoplasm most commonly diagnosed in both sexes and the second leading cause of cancer death in Spain. Colorectal cancer screening Program in Barcelona was implanted in 2009 and approximately 1,500 colorectal cancer screening colonoscopies are performed annually at Hospital Clínic de Barcelona. Adequate colon preparation (anterograde cleansing with laxatives) improves polyp detection, decreases examination time, and complications. There are both low and high volume intestinal regimens with polyethylene glycol (PEG) as the main active ingredient or without it.

Hypothesis: Two low volumen regimens, 1L PEG plus ascorbate and magnesium citrate plus picosulphate, at starting doses have the same Adenoma Detection Rate as cleansing solutions in preparation for screening colonoscopy.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the clinical efficacy (by comparing the adenoma detection rate) of 1L PEG plus ascorbate versus magnesium citrate plus picosulphate in subjects undergoing colonoscopy in a colorectal cancer screening programme. We also will compare the Lesion Detection Rate, the quality of colon cleansing (Boston classification) overall and by segments, the tolerability and satisfaction and the rate of adverse effects experienced with intake of these products.

Methodology: A comparative, parallel, randomized, single-centre, low-intervention clinical trial to be conducted at the CCR screening unit of Hospital Clínic de Barcelona that will include 1,002 participants.

Subjects will complete a Tolerability and Satisfaction Questionnaire after completing the bowel preparation. Findings (polyps, CRC, or other lesions) and quality of bowel cleansing will be collected from the colonoscopy report.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50 to 69 years who have participated in the early detection programme for colon and rectal cancer (PDPCCR) in Barcelona, who have obtained a positive result in the faecal occult blood test (≥20 μg Hb/g faeces) and who are scheduled for a screening colonoscopy at Hospital Clínic de Barcelona.

Exclusion Criteria:

* People who do not agree to participate in the study.
* People with known severe renal failure (grade IV or V) and grade III and IV heart failure according to the New York Heart Association (NYHA) Scale of Functional Assessment of Heart Failure
* Individuals who have undergone a colonoscopy in the past year.
* Subjects meeting the Rome IV Criteria for the diagnosis of functional constipation
* Subjects with mental disabilities or with a severe mental disorder (schizophrenia and other psychotic disorders, recurrent severe major depressive disorders, severe obsessive-compulsive disorder, severe personality disorders and bipolar disorders).
* Individuals who do not understand Catalan or Spanish verbally and in writing.
* Individuals with partial or total colon resection.
* Individuals with a personal history of CRC or colorectal disease amenable to specific follow-up (ulcerative colitis, Crohn's disease, or colorectal adenomas).
* Individuals with terminal illness or severe illness/disability that contraindicates further study of the colon.
* People with gastrointestinal disorders that contraindicate the use of the study products (gastric emptying disorders, perforation or gastrointestinal obstruction, ileus, toxic megacolon).
* People with congestive heart failure
* Hypermagnesemia
* Rhabdomyolysis
* Phenylketourine
* Glucose-6-phosphate dehydrogenase deficiency
* People with hypersensitivity to the active ingredients of excipients
* People with severe renal impairment

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 2 years
  The percentage of patients with at least one adenoma in relation to the total subjects in each group of study

SECONDARY OUTCOMES:
Colonoscopy quality | 2 years
  Colonoscopy quality is assess with Boston Bowel Preparation Scale (BBPS) in which each colon segment (right colon, transverse colon, and left colon) is scored from 0 to 3 (0=poor, 1=fair, 2=good, 3=excellent). It will be considered adequate when each segment is scored ≥2.
Lesion detection rate | 2 years
  The percentage of patients with at least one polyp in relation to the total subjects in each group
Caecal intubation rate | 2 years
  If the caecum has been reached in the colonoscopy, it will be considered complete; otherwise, it will be considered incomplete
Rate of adverse events related to the administration of the preparation | 2 years
  Evaluated with the Tolerability and Satisfaction Questionnaire including symptoms such as nausea, vomiting, abdominal pain, bloating, headache, chills, dizziness, and dry mouth
Tolerability and satisfaction with preparation | 2 years
  Assessed by completing a tolerability and satisfaction questionnaire that has been prepared from the validated questionnaire Mayo Clinic Bowel Prep Tolerability Questionnaire (Patel M, Staggs E, Thomas CS, Lukens F, Wallace M, Almansa C. Development and validation of the Mayo Clinic Bowel Prep Tolerability Questionnaire. Dig Liver Dis. 2014 Sep; 46(9):808-12.doi: 10.1016/j.dld.2014.05.020. Epub 2014 Jun 19. PubMed PMID: 24953203) and which has been adapted and translated into Spanish

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital CLinic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hautefeuille G, Lapuelle J, Chaussade S, Ponchon T, Molard BR, Coulom P, Laugier R, Henri F, Cadiot G. Factors related to bowel cleansing failure before colonoscopy: Results of the PACOME study. United European Gastroenterol J. 2014 Feb;2(1):22-9. doi: 10.1177/2050640613518200. PMID 24918005
- [Background] Schreiber S, Baumgart DC, Drenth JPH, Filip RS, Clayton LB, Hylands K, Repici A, Hassan C; DAYB Study Group. Colon cleansing efficacy and safety with 1 L NER1006 versus sodium picosulfate with magnesium citrate: a randomized phase 3 trial. Endoscopy. 2019 Jan;51(1):73-84. doi: 10.1055/a-0639-5070. Epub 2018 Jul 19. PMID 30025415
- [Background] Bisschops R, Manning J, Clayton LB, Ng Kwet Shing R, Alvarez-Gonzalez M; MORA Study Group. Colon cleansing efficacy and safety with 1 L NER1006 versus 2 L polyethylene glycol + ascorbate: a randomized phase 3 trial. Endoscopy. 2019 Jan;51(1):60-72. doi: 10.1055/a-0638-8125. Epub 2018 Jul 19. PMID 30025414
- [Background] DeMicco MP, Clayton LB, Pilot J, Epstein MS; NOCT Study Group. Novel 1 L polyethylene glycol-based bowel preparation NER1006 for overall and right-sided colon cleansing: a randomized controlled phase 3 trial versus trisulfate. Gastrointest Endosc. 2018 Mar;87(3):677-687.e3. doi: 10.1016/j.gie.2017.07.047. Epub 2017 Aug 10. PMID 28803744
- [Background] Seo SI, Kang JG, Kim HS, Jang MK, Kim HY, Shin WG. Efficacy and tolerability of 2-L polyethylene glycol with ascorbic acid versus sodium picosulfate with magnesium citrate: a randomized controlled trial. Int J Colorectal Dis. 2018 May;33(5):541-548. doi: 10.1007/s00384-018-2989-7. Epub 2018 Mar 1. PMID 29497812
- [Background] Lee SW, Bang CS, Park TY, Suk KT, Baik GH, Kim DJ. Split-dose Bowel Preparation for Colonoscopy: 2 Liters Polyethylene Glycol with Ascorbic Acid versus Sodium Picosulfate versus Oral Sodium Phosphate Tablets. Korean J Gastroenterol. 2017 Aug 25;70(2):89-95. doi: 10.4166/kjg.2017.70.2.89. PMID 28830134
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Patel M, Staggs E, Thomas CS, Lukens F, Wallace M, Almansa C. Development and validation of the Mayo Clinic Bowel Prep Tolerability Questionnaire. Dig Liver Dis. 2014 Sep;46(9):808-12. doi: 10.1016/j.dld.2014.05.020. Epub 2014 Jun 19. PMID 24953203
- [Background] Guillaumes S, O'Callaghan CA. [Spanish adaptation of the free OxMaR software for minimization and randomization of clinical studies]. Gac Sanit. 2019 Jul-Aug;33(4):395-397. doi: 10.1016/j.gaceta.2018.07.013. Epub 2018 Nov 1. Spanish. PMID 30390995
- See also: Las cifras del cáncer en España 2018 - SEOM: Sociedad Española de Oncología Médica © 2019 — https://seom.org/ultimas-noticias/106525-las-cifras-del-cancer-en-espana-2018.
- See also: Guía clínica de Calidad en la Colonoscopia de Cribado del CCR — http://www.aegastro.es/publicaciones/publicaciones-aeg/guias-de-practica-clinica/guia-clinica-de-calidad-en-la-colonoscopia-de-cribado-del-cancer-colorrectal